CLINICAL TRIAL: NCT01078285
Title: Impact Of An Integrated Intervention Program On Adherence To Atorvastatin
Brief Title: Effectiveness Of A Program That Includes Counseling And Patient Support On Adherence To Treatment With Lipitor
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A2581184
Record Dates: First submitted 2010-02-25; First posted 2010-03-02 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Medication Non-Adherence
Keywords: Integrated program on adherence using counseling; support services including cost-sharing where appropriate and educational materials mailed monthly.
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control
  Interventions: Behavioral: No Patient Counseling
- Intervention Arm
  Interventions: Behavioral: Adherence Counseling

INTERVENTIONS:
Behavioral: No Patient Counseling — Patients do not receive any adherence counseling, or other patient support services
  Groups: Control
Behavioral: Adherence Counseling — Patients receive 3-5 minutes of adherence counseling, and other patient support services
  Groups: Intervention Arm

SUMMARY:
Despite extensive reports of the benefits of statins in reducing serious cardiovascular events such as stroke and heart disease in patients with elevated LDL-cholesterol, patients do not take their medicines regularly as prescribed. Reasons include forgetfulness, lack of understanding of the seriousness of the disease, and fear of side effects. An intervention strategy comprising 3-5 minutes of counseling, emotional support and cost-sharing may be motivational and improve adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged >21 years
* Have received a new or re-fil prescription for atorvastatin at first study visit to Prairie Heart Institute
* Signed informed consent

Exclusion Criteria:

* Unwilling to give written informed consent
* Failed statin treatment in the past
* Switched from another statin to atorvastatin because of co-pay program
* Participated in an earlier Market Research study on Impact of cholesterol management behaviors post in-clinic adherence intervention

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Male and female aged >21 years
  * Have received a new or re-fil prescription for atorvastatin at first study visit to Prairie Heart Institute
  * Signed informed consent
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Proportion of Days Covered (PDC) | 180 days

SECONDARY OUTCOMES:
Medication Possession Ratio (MPR) | 180 days
Persistence-the number of continuous days a patient is supplied with medication using the allowable grace period or gap (30 or 60 days). | 180 days
Percent of patients that are at least 80% adherent (PDC>0.8) | 180 days
Percent of patients who fill at least one atorvastatin prescription during the period of study | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Prairie Heart Institute, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Prairie Diagnostic Center, Springfield, Illinois

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581184&StudyName=Effectiveness%20Of%20A%20Program%20That%20Includes%20Counseling%20And%20Patient%20Support%20On%20Adherence%20To%20Treatment%20With%20Lipitor